CLINICAL TRIAL: NCT01380054
Title: Pulmonary Hypertension: Impact of the Evolution of a Rare Disease on the Quality of Life and Role of Variables Psychosocial as Predictive of the Current and Later Quality of Life
Brief Title: Pulmonary Hypertension, Quality of Life and Psychosocial Factors
Acronym: HyPsy
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 8705; 2011-A00174-37 (Other: AFSSAPS)
Record Dates: First submitted 2011-06-06; First posted 2011-06-27 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Quality of life; Coping; Depression; Anxiety; Social support; Control beliefs
MeSH Terms: conditions — Hypertension, Pulmonary; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with pulmonary hypertension
  Interventions: Behavioral: Evaluation of quality of life

INTERVENTIONS:
Behavioral: Evaluation of quality of life — -Psychological interviews-Questionaires : HAD, STAI, CHIP, MHLC, WCC, SSQ scales-Quality of life : SF-36

SUMMARY:
The investigators aim to :

* describe and analyse psychological characteristics, cognitive factors and representations in patients with Pulmonary Hypertension, a rare disease.
* assess the psychological characteristics impact on quality of life, check the association between disease and QoL evolution, and the variability of QoL parameters over severity class changes and follow-up

DETAILED DESCRIPTION:
PAH is a rare, and severe disease, potentially mortal, affecting preferentially young subjects. The knowledge and the international literature, as regards the quality of life, the expectations, the needs and the psychosocial characteristics of patients with PAH, are non-existent. But it is known that the persons affected by rare diseases are more vulnerable, on the psychological, social, economic and cultural planIn all the stages of the treatment, patients with PAH are confronted with heavy psychosocial situations, in a context of vital risk, with exceptional medicinal treatments (intravenous administration at home).

* QoL might be differently affected by these changes according to situational and dispositional psychological dimensions.
* the predictive role of these characteristics on the current and later quality of life, as well as the impact of diverse cognitive mediators and strategies to cope with the disease, should be investigated.The respiratory diseases department of the Montpellier hospital is regional competence center for PAH in Languedoc-Roussillon, under the aegis of the national reference center (the respiratory diseases department of Antoine Béclère hospital, Le Petit-Clamart).

ELIGIBILITY:
Inclusion Criteria:

* Patients with PAH
* Patients stable since 3 months
* Patients with a severity of class I to IV
* Patients aged between 18 and 80 years
* Patients no psychological follow-up at the competence center.

Exclusion Criteria:

* Patients unable to give his accordance
* Patients unable to understand the aim of the study
* Patients with recents psychiatrics disorders
* Patients with problems of understanding the tests of the study
* Drug users or drinkers
* Pregnant or women without efficacy contraception
* Patient without freedom by administration decision
* Patient in exclusion period
* Patient without french insurance
* Adult protected by the law

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PAH, aged between 18 and 80 years, stable since 3 months, no psychological follow-up at the competence center.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2011-05-31 (Actual); Primary Completion 2016-05-20 (Actual); Study Completion 2016-05-20 (Actual)

PRIMARY OUTCOMES:
Descriptive analysis of psychological characteristics on PAH patients | 36 months
  The descriptive analysis of psychological characteristics (anxiety, depression, social support, coping, control beliefs) is evaluated at entry and at one year. These psychological characteristics are evaluated by score of psychological questionnaires.

SECONDARY OUTCOMES:
Psychological characteristics impact on Quality of life | 36 months
  The quality of life is measured by the score of the SF 36, the stage of the disease is codified by the NYHA, Qualitative and quantitative analysis of contents of the audio bands by the psychologist implicated to this study.
Association between disease and Quality of life evolution | 36 months
  The quality of life is measured by the score of the SF 36, the stage of the disease is codified by the NYHA, Qualitative and quantitative analysis of contents of the audio bands by the psychologist implicated to this study.
Variability of Quality of life parameters over severity class changes and follow-up | 36 months
  The quality of life is measured by the score of the SF 36, the stage of the disease is codified by the NYHA, Qualitative and quantitative analysis of contents of the audio bands by the psychologist implicated to this study.

CONTACTS AND LOCATIONS:
Overall Officials: Bourdin Arnaud, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- CHU, Montpellier, France

REFERENCES:
- [Result] Halimi L, Suehs CM, Marin G, Boissin C, Gamez AS, Vachier I, Molinari N, Bourdin A. Health-related quality of life and disease progression in pulmonary arterial hypertension patients: a 3-year study. ERJ Open Res. 2021 Aug 23;7(3):00617-2020. doi: 10.1183/23120541.00617-2020. eCollection 2021 Jul. PMID 34435036
- [Result] Halimi L, Marin G, Molinari N, Gamez AS, Boissin C, Suehs CM, Vachier I, Bourdin A. Impact of psychological factors on the health-related quality of life of patients treated for pulmonary arterial hypertension. J Psychosom Res. 2018 Feb;105:45-51. doi: 10.1016/j.jpsychores.2017.12.003. Epub 2017 Dec 6. PMID 29332633
- See also: HyPsy on the Open Science Framework. — http://osf.io/8qduc